CLINICAL TRIAL: NCT05202171
Title: The Effects of Cervical Stabilization Exercise Training With Telerehabilitation in Individuals With Migraine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, seyda toprak celenay, associate professor, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/01/8
Record Dates: First submitted 2022-01-10; First posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Exercise group will be performed cervical stabilization exercise training applied with telerehabilitation and standard treatment ( preventive/symptomatic oral drug therapy routinely in the clinic and suggestions for triggering factors in migraine) for 8 weeks
  Interventions: Other: Cervical Stabilization Exercise
- Standard treatment group (Active Comparator): Standard treatment group will be given preventive/symptomatic oral drug therapy routinely in the clinic and suggestions for triggering factors in migraine for 8 weeks.
  Interventions: Other: Standard treatment

INTERVENTIONS:
Other: Cervical Stabilization Exercise — Exercise group will be performed cervical stabilization exercise training applied with telerehabilitation and standard treatment ( preventive/symptomatic oral drug therapy routinely in the clinic and suggestions for triggering factors in migraine) for 8 weeks
  Arms: Exercise group
Other: Standard treatment — standard treatment will include preventive/symptomatic oral drug therapy routinely in the clinic and suggestions for triggering factors in migraine for 8 weeks
  Arms: Standard treatment group

SUMMARY:
The aim of our study is to investigate the effects of cervical stabilization exercise training applied with telerehabilitation in individuals with migraine.

DETAILED DESCRIPTION:
Cervical muscles are adversely affected in individuals with migraine. It is important to investigate the effects of cervical muscle training in these individuals. Telerehabilitation applications have been used frequently in many patients in recent years. It is necessary to examine the effects of cervical stabilization exercises applied with telerehabilitation in individuals with migraine.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-55,
* To be diagnosed with migraine by a neurologist according to International Headache Society criteria,
* Having at least 3 migraine attacks per month,
* Volunteering to participate in the study,
* Having the opportunity to access devices such as computers, phones and tablets with internet connection,
* Not having any problems that prevent cooperation and understanding

Exclusion Criteria:

* Having other accompanying headache types,
* Being pregnant,
* Being in the breastfeeding period,
* Having a history of trauma, fracture or surgery in the craniocervical region,
* Presence of concomitant neurological and/or inflammatory rheumatic disease
* Presence of serious psychiatric problems,
* History of malignancy,
* Changes in medical treatment during the study period,
* Receiving physiotherapy for the cervical region in the last 6 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
The characteristic of the migraine | change from baseline at 8 weeks
  The characteristic of the migraine will be evaluated with the "Headache Diary".

SECONDARY OUTCOMES:
Cervical range of motion | change from baseline at 8 weeks
  Cervical range of motion was evaluated using the goniometer
Upper cervical region movements | change from baseline at 8 weeks
  Upper cervical region movements will be evaluated with a Cervical Range of Motion device
Performance of the deep neck flexor muscles | change from baseline at 8 weeks
  Performance of the deep neck flexor muscles will be evaluated with a Stabilizer Pressure Biofeedback Unit
Cranio-vertebral angle | change from baseline at 8 weeks
  The cranio-vertebral angle will be measured with a goniometer
Disability Status | change from baseline at 8 weeks
  The Turkish version of Migraine Disability Assessment Scale will be used to determine the disability status in daily activities of individuals due to migraine
Sleep quality | change from baseline at 8 weeks
  Sleep quality will be evaluated with the Turkish version of Jenkins Sleep Scale
Life quality | change from baseline at 8 weeks
  Life quality will be evaluated with the Turkish version of Headache Impact Test

CONTACTS AND LOCATIONS:
Overall Officials: Seyda Toprak Celenay, Principal Investigator — Ankara Yildirim Beyazıt University